CLINICAL TRIAL: NCT06327438
Title: Complex Decongestive Therapy, Cryotherapy and Kinesio Taping in Patients With Post-mastectomy Lymphedema
Brief Title: Effect of Complex Decongestive Therapy, Cryotherapy and Kinesio Taping in Patients With Post-mastectomy Lymphedema: A Randomized Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Ragaee Saeed Mahmoud, Lecturer, National Cancer Institute (NCI)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/211/MTI.PT/2401041
Record Dates: First submitted 2024-03-15; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Breast Neoplasms
Keywords: Complex Decongestive Therapy; Cryotherapy; Kinesio Taping; Lymphedema; Post-mastectomy
MeSH Terms: conditions — Breast Neoplasms; Lymphedema | interventions — Cryotherapy

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A) (Experimental): (n=20) received complex decongestive therapy only
  Interventions: Other: Complex decongestive therapy
- Group (B) (Experimental): (n=20) received cryotherapy and complex decongestive therapy
  Interventions: Other: Complex decongestive therapy; Device: Cryotherapy
- Group (C) (Experimental): (n=20) received kinesio taping and complex decongestive therapy
  Interventions: Other: Complex decongestive therapy; Other: Kinesio taping

INTERVENTIONS:
Other: Complex decongestive therapy — 1. Manual lymphatic drainage (MLD).
  2. Compression bandage.
  3. Exercises to enhance lymphatic drainage.
  4. Skin care.
Device: Cryotherapy — It is a mature and safe-to-use system that cools the air to -32°C. Steps of application included: 1) Apply oil or cream to moisture the skin before cryotherapy application; 2) Initialize the mini cryo-air equipment at level 6.
  Arms: Group (B)
Other: Kinesio taping — It is a new choice in the field of physical therapy. The material used for the KT and the original concept of the taping technique were introduced by Dr Kenso Kase in 1973.
  Arms: Group (C)

SUMMARY:
To examine the efficacy of complex decongestive therapy (CDT), cryotherapy and kinesio taping (KT) in patients with post-mastectomy lymphedema

DETAILED DESCRIPTION:
Sixty women diagnosed clinically by physician as post-mastectomy lymphedema, suffered from grade 2 and 3 lymphedema based on clinical investigations and their ages between 40 and 60 years were randomly assigned in single pre - post measurement study. They divided randomly into three groups of equal size (A, B & C). The three groups received CDT program, group (A) (n=20) received CDT only, group (B) (n=20) received cryotherapy and group (C) (n=20) received KT

ELIGIBILITY:
Inclusion Criteria:

Patients aged between 40 to 60 years. They were grade 2 and 3 lymphedema. They had more than 2 cm difference at circumference measurement. They had unilateral arm lymphedema post-mastectomy. They had completed chemotherapy and radiotherapy.

Exclusion Criteria:

Skin infection. Current ischemia. Systemic edema due to impaired heart, kidney and liver function. Current metastases. Venous thrombosis.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-16 (Estimated); Primary Completion 2024-06-16 (Estimated); Study Completion 2024-07-16 (Estimated)

PRIMARY OUTCOMES:
Arm girth measurement is measured by Circumferential measurements | 12 consecutive weeks
  It is a valid and reliable method, its protocol was used throughout, with measures performed on both arms at the axilla, halfway from the axilla to the cubital fossa, cubital fossa, halfway from the cubital fossa to the wrist, and at the wrist.
Pain severity is measured by VAS | 12 consecutive weeks
  It consisted of a line, often 10 cm long (100 mm); its ends are generally labelled with verbal pain anchors (e.g., "no pain" and "pain as bad as it could be")

SECONDARY OUTCOMES:
The QOL is measured by SF-36 | 12 consecutive weeks
  It is widely validated and popularly method that is used to evaluate QOL of the patients. Since then, the reliability and validity of the SF-36 questionnaire have been evaluated in a number of specific population world-wide
Range of motion (ROM) is measured by UG | 12 consecutive weeks
  It is GONIO_PLASTIC_360, China, frequently used for measurement of shoulder ROM (flexion, abduction and external rotation) by physical therapists to assess ROM due to its ease of use, portability, noninvasive nature, and low cost

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ragaee Saeed Mahmoud, Giza, Faisal
  - Ragaee Saeed Mahmoud, Faisal, Giza Governorate

IPD SHARING:
Plan to Share IPD: No
Intervention